CLINICAL TRIAL: NCT01575743
Title: Effects of Aerobic Exercise on Occupational Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Burnout_1
Record Dates: First submitted 2012-04-03; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Burnout Syndrome
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: aerobic exercising
- healthy controls (Other)
  Interventions: Behavioral: aerobic exercising

INTERVENTIONS:
Behavioral: aerobic exercising — All participants take part in an aerobic exercise training program with a total weekly energy expenditure of 17.5 kcal/kg/week over the entire 12-week intervention period. The dose of exercise is determined using exercise prescription guidelines established by the American College of Sports Medicine (ACSM, American College of Sports Medicine, 2000). All trainings take place at a local public gym under supervision of previously trained exercise coaches from the Institute of Exercise and Health Sciences of the University Basel. Participants can choose between different training devices for cardiovascular training. Energy expenditure is assessed using the values of burned calories provided by the training devices based on age, weight and training performance. Heart rate is monitored during all training sessions with chest belt heart rate monitors (Polar®) to ensure training below the anaerobic threshold with heart rates between 60 - 75 % of the maximum heart rate.

SUMMARY:
The aim of the present study is to investigate the impact of regular aerobic exercise on psychopathology, cortisol secretion, BDNF, sleep, cognitive performance, and psychological functioning in people suffering from professional burnout. Pre- and postassessments after 12 weeks of training will be performed.

ELIGIBILITY:
Inclusion Criteria:

* burnout
* male participants
* non-smokers

Exclusion Criteria:

* psychiatric disorders
* smokers
* physical diseases

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change of burnout severity by aerobic exercise training | Change from baseline to follow-up after 12 weeks
  burnout severity measured by psychopathology, cortisol secretion, BDNF, sleep, cognitive performance, and psychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Beck, MD, Principal Investigator — UPK Basel, Basel Switzerland
Locations (1):
- UPK Basel, Basel, Switzerland, Switzerland

REFERENCES:
- [Derived] Gerber M, Brand S, Elliot C, Holsboer-Trachsler E, Puhse U, Beck J. Aerobic exercise training and burnout: a pilot study with male participants suffering from burnout. BMC Res Notes. 2013 Mar 4;6:78. doi: 10.1186/1756-0500-6-78. PMID 23497731